# Pancreatic Enzyme Replacement Therapy for treatment of Exocrine Pancreatic Insufficiency in Patients with Unresectable Pancreatic Cancer

NCT02985801

May 15, 2018

### **IRB Minimal Risk Protocol Template**

Note: If this study establishes a human specimen repository (biobank) for research purposes, do not use this template. Use the Mayo Clinic Human Specimen Repository Protocol Template found on the IRB home page under Forms and Procedures at http://intranet.mayo.edu/charlie/irb/

**First-time Use:** Use this template to describe your study for a new IRB submission.

- 1. Complete the questions that apply to your study.
- 2. Save an electronic copy of this protocol for future revisions.
- 3. When completing your IRBe application, you will be asked to upload this template to the protocol section.

**Modification:** To modify this template <u>after</u> your study has been approved:

- 1. Open your study in IRBe. Click on the study 'Documents' tab and select the most recent version of the protocol. Save it to your files.
- 2. Open the saved document and activate "Track Changes".
- 3. Revise the protocol template to reflect the modification points, save the template to your files
- 4. Create an IRBe Modification for the study and upload the revised protocol template.

# **General Study Information**

Principal Investigator: Massimo Raimondo, M.D.

Study Title: Pancreatic Enzyme Replacement Therapy for treatment of Exocrine Pancreatic Insufficiency in Patients with Unresectable Pancreatic Cancer

Protocol version number and date: version 5, 5/15/2018

# **Purpose**

#### Hypothesis:

Pancreas enzyme replacement therapy (PERT) decreases weight loss and improves quality of life in patients with unresectable pancreatic cancer.

Aims, purpose, or objectives:

- 1. Assess prevalence of pancreatic exocrine insufficiency (PEI) with fecal elastase-1 test (FE1) in patients with unresectable pancreatic cancer, without evidence of pancreatic duct (PD) or common bile duct (CBD) obstruction based on MRI or / and EUS.
- 2. Patients with PEI (FE1 <200) receive Pertzye or placebo in a cross-over fashion, each for 4 weeks. 3 capsules are taken with or after meals and 2 capsules with or after snacks (approximating 500 lipase units/kg/meal).

- 3. Body weight, body mass index (BMI), body composition (Bodystat Bioimpedance), are measured at the time of diagnosis of PEI and at 4 and 8 weeks of cross-over treatment. Baseline measurement of Vitamin D-25, Vitamin A, iron (ferritin, TIBC, iron), Vitamin B12, Tissue transglutaminase IgA (tTG) with total Immunoglobulin A (IgA)
- 4. Quality of Life (pain, diarrhea, weight, bloating, etc.) assessed at 0,4,8 weeks with

a.

b. Functional Assessment (FACT-Hep) for physical, social, emotional, and functional QOL<sup>2</sup>

# Background

Pancreatic exocrine insufficiency (PEI) is a known complication of pancreatic cancer. Several mechanisms of PEI have been described in context of pancreatic cancer, including pancreatic atrophy secondary to tumor induced pancreatic duct obstruction and pancreatic fibrosis, both leading to PEI in patients with unresectable pancreatic cancer.<sup>3</sup>

Although the majority of patients with pancreatic cancer are inoperable at the time of diagnosis, only few authors addressed PEI in this patient cohort. Small studies with 8 to 12 patients detected PEI in 75% to 100%. The prevalence of PEI tended to be higher in setting of significant pancreatic duct obstruction. <sup>4,5</sup> The largest cohort study included 194 patients with advanced pancreatic cancer which was defined as metastatic or unresectable due to local invasion. 50% of study participants had PEI. As a next step, Sikkens et al prospectively assessed the progression of PEI in 32 patients with unresectable cancer of the pancreatic head region. Based on FE1 testing, 67% of patients had PEI at the time of pancreatic cancer diagnosis and 89% at 2 months follow up (median).

Despite a high prevalence of PEI in patients with unresectable pancreatic cancer, clinical symptoms like steatorrhea are not uniformly present. In fact, 2 hallmark studies, including one with 12 and one with 194 patients, found no statistically significant correlation between the dyspepsia, number of bowel movements on the one hand and the presence of fat malabsorption on the other hand in patients with unresectable pancreatic cancer. Only 16.7% of patients with very severe PEI had clinically evident steatorrhea, whereas 5.2% of patients had subjective steatorrhea without PEI.<sup>5,6</sup> Weight loss is another well-known complication of pancreatic cancer. Perez et al. who found a significant correlation between fat-protein malabsorption and weight loss in non-surgical patients with pancreatic cancer however not between diminished caloric consumption and weight loss.<sup>5</sup>

As of now, multiple studies showed improved fat absorption with pH-sensitive microsphere formulation in comparison to conventional pancreatic enzyme preparations or placebo in chronic pancreatitis patients with PEI.<sup>8-14</sup> However, only few studies addressed the utility of PERT for patients with inoperable pancreatic cancer, including a randomized study by Bruno et al. with 21 patients with unresectable pancreatic cancer and pancreatic duct obstruction. Patients randomized into PERT for 4 weeks had reduced weight loss compared with patients who were treated with placebo.<sup>15</sup> A retrospective study by Domínguez-Muñoz et al. included 76 patients with inoperable pancreatic cancer. Patients who received PERT (Creon<sup>®</sup>) had a longer median survival than patients with palliative therapy alone.<sup>16</sup> Of note, PEI was not formally assessed in either of those studies. Based on these limited results current pancreatic cancer guidelines recommend PERT for patients with unresectable pancreatic cancer, in the realm of palliative therapy.<sup>17</sup> However the efficacy of PERT in patients with unresectable pancreatic cancer was never proven in a randomized controlled trial.

A further concern is the adverse drug reaction profile of PERT. In adult population no severe side effects of PERT are documented. Hyperuricosuria and especially colonic fibrosis are the most feared severe adverse drug reaction (ADR) of long term PERT, however they were reported only in children with cystic fibrosis. <sup>18,19, 20,21</sup>

However dyspepsia, heartburn and bloating are well described mild ADR of PERT. In this context, several randomized controlled trials revealed a higher incidence of bloating and abdominal pain in patients who received PERT for PEI for mostly benign pancreatic conditions. <sup>21,22,23,24</sup> The impact of ADR on the quality of life was never assessed in a randomized controlled fashion in patients with unresectable pancreatic cancer. Finally, the high costs of PERT, which range up to \$2000 a month, emphasis the importance to clarify the pros and cons of PERT for patients with unresectable pancreatic cancer, to avoid unnecessary and costly treatments.

# Subject Information – charts, records, images, or specimens are considered 'subjects'

Target accrual is the proposed number of subjects to be included in your study at your site. "Subjects" may include Mayo Clinic charts, records, or specimens, **and/or** charts, records, or specimens received at Mayo Clinic from external sources for collaborating analysis by the investigator under this IRB application:

Target accrual:

30 completed patients

Subject population:

#### **Inclusion Criteria:**

- Patients 18- 100 years
- Underlying pancreatic adenocarcinoma, unresectable (local invasion or distant metastasis)
- On established chemotherapy regimen for pancreas cancer, which will be continued over the time of study
- Fecal elastase-1 test (FE1) less than 200 mcg pancreatic elastase/g stool

#### **Exclusion Criteria:**

- Common bile duct obstruction resulting in obstructive jaundice
- Celiac disease
- Crohn's disease
- Benign pancreatic conditions
- Bowel obstruction
- Surgically altered bowel anatomy

| Yes No Will a Certificate of Confidentiality (COC) be obtained from NIH? If yes, |
|---|
| Who is obtaining the COC: Mayo Clinic investigator, study sponsor, other: |
| Explain why a COC is needed: |
| Study Design |

#### Methods:

Patients with unresectable pancreatic adenocarcinoma (local invasion or distant metastasis) receive pancreatic enzyme replacement therapy (PERT) by the oncology team as presumed standard of care. Patients will be offered to participate in study, which lasts 10 weeks.

Pancreatic enzyme insufficiency (PEI) will be detected by (fecal elastase-1) FE1 testing. Patients with FE1 less than 200 mcg pancreatic elastase/g stool are eligible for study. Patients will be randomized into first placebo or first treatment group (cross over study) by enclosed envelope.

Patients will received either Pertzye (Pancrelipase) 500 lipase units/kg/meal or placebo, each for 4 weeks. Dosing will be 3 capsules 3 times a day with or after meals and 2 capsules with or after snacks. No treatment will be administered at weeks 5 and 6 to assure adequate washout. Pertzye or placebo will be given for another 4 weeks (week 7 - 10) in a cross-over fashion.

Body weight, body mass index (BMI), body composition (Tanita, TBF-310GS, Bodystat Bioimpedance), FACT-Hep quality of life assessment will be measured at randomization and at last day of treatment or placebo (week 4 and 10).

#### Resources:

Patients will be recruited in oncology or gastroenterology clinic by oncology fellow or gastroenterology fellow in the setting of their regular clinical work.

Pertzye and placebo will be sponsored by pharmaceutical company.

# Check all that apply. If none apply, leave blank:

| This is a multisite study involving Mayo Clinic and non-Mayo Clinic sites. When checked, describe the research procedures/activities being conducted <b>only</b> at Mayo Clinic: |
|---|
| Mayo Clinic staff will be engaged in research activity at a non-Mayo Clinic site. When checked, provide the location and a detailed description of the Mayo Clinic research staff involvement. |
| ☐ This study is to establish and/or maintain an ongoing database or registry for research purposes only. |
| ☐ The research involves contact or interaction with subjects, for example, surveys, questionnaires, observation, blood draw. |
| ☐ The study involves photographing, audiotaping or videotaping subjects (and guests). |
| Review of Chart, Images, Specimens |
| Provide the date range for collection of data and/or specimens that will be included in your research dataset. |
| Check all that apply: |
| This study involves only data and/or specimens that exist at the time this application is submitted to the IRB (IRB submission date). No data or specimens will be collected beyond this date. |

| Data Confidentiality, HIPAA Subject Identifiers |
|---|
| Other data sources will be utilized in this study, e.g. receiving data/specimens from an external party. When checked, provide all data sources: |
| Note: When subjects provided consent for use of their data and/or specimens, as described in this protocol. |
| IRB Number/s - Data and Specimens: |
| IRB Number/s - Specimens Only: |
| IRB Number/s - Data Only: |
| Data and/or specimens used in this study are collected under another IRB protocol. When checked, provide the IRB number(s) from which the research material will be obtained. When appropriate, check the box below to attest that subjects have provided consent for future use of their data and/or specimens, as described in this protocol. |
| The study involves data and/or specimens that exist at the time of submission to the IRB <u>and</u> data and/or specimens that will be collected after submission to the IRB, for example a study that includes collection of existing data and prospective collection of specimens. |
| x This study involves only data and/or specimens that will be collected after submission to the IRB. |

Review the list of subject identifiers below and, if applicable, check the box next to each subject identifier being recorded at the time you are collecting/abstracting data/specimens for use in this study.

**Subject Identifiers**: Individually identifiable information, including demographic data, that identifies the individual or for which there is reasonable basis to believe it can be used to identify the individual. NOTE: Identifiers apply to subjects enrolled in your study and to the subject's relatives, household members, employers, etc.

**Internal** refers to subject identifiers that will be included in the dataset maintained by the study team. **External** refers to subject identifiers that will be shared with persons outside of the immediate study team, for example, sent to an external collaborator or shared with a national registry.

| SUBJECT IDENTIFIERS Check all that apply | INTERNAL<br>IDENTIFIER | EXTERNAL IDENTIFIER |
|---|---|---|
| Name | X | |
| Social Security number | | |
| Medical record/patient registration number, lab accession, specimen or | X | |
| radiologic image number | | |

| Study number, subject ID, or any other unique identifying number, | X | |
|---|---|---|
| characteristic or code that can be used to link the identity of the subject to the | | |
| data | | |
| Dates: All elements of dates [month, day, and year] directly related to an | X | |
| individual. Their birth date, date of death, date of diagnosis, etc. | | |
| <b>Note:</b> Recording a year only is not a unique identifier. | | |
| Medical device identifiers and serial numbers | | |
| Biometric identifiers, including finger and voice prints, full face photographic | | |
| images and any comparable images | | |
| Web Universal Resource Locators (URLs), Internet Protocol (IP) address | | |
| numbers, email address | | |
| Street address, city, county, precinct, zip code, and their equivalent geocodes | | |
| Phone or fax numbers | | |
| Account, member, certificate or professional license numbers, health | | |
| beneficiary numbers | | |
| Vehicle identifiers and serial numbers, including license plate numbers | | |
| If None of the above identifiers will be recorded or maintained in the | None | None |
| dataset and/or sent outside of the study team, please check "None". | ∐ None | ∐ None |

# **Statistical Information**

# **Statistical Considerations**

Data Analysis Plan and Power Statement:

Statistical significance will be calculated with pair t-test.

According to Bruno et al and Dominguez-Munoz et al a 5% weight difference between the treatment groups is expected within 4 weeks. Standard deviation is expected to be less than 5% based on the cross over fashion. Assuming a patient drop out of 30%, a minimum of 13 patients need to be included in the trial to detect a statistically significant difference, with a power of 80% and alpha error of 5%. Eventually, we target to include 30 patients to assure adequate power, given the statistical limitations of previously reviewed studies.

# **Endpoints**

# Primary:

1. Weight change

# Secondary:

- 1. Quality of life (QOL)
- 2. Change in body composition

#### References

- 1. Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. The British journal of surgery 1995;82:216-22.
- 2. Heffernan N, Cella D, Webster K, Odom L, Martone M, Passik S, Bookbinder M, Fong Y, Jarnagin W, Blumgart L. Measuring health-related quality of life in patients with hepatobiliary cancers: the functional assessment of cancer therapy-hepatobiliary questionnaire. Journal of clinical oncology: official journal of the American Society of Clinical Oncology 2002;20:2229-39.
- 3. Ghaneh P, Neoptolemos JP. Exocrine pancreatic function following pancreatectomy. Annals of the New York Academy of Sciences 1999;880:308-18.
- 4. DiMagno EP, Malagelada JR, Go VL. The relationships between pancreatic ductal obstruction and pancreatic secretion in man. Mayo Clinic proceedings 1979;54:157-62.
- 5. Perez MM, Newcomer AD, Moertel CG, Go VL, Dimagno EP. Assessment of weight loss, food intake, fat metabolism, malabsorption, and treatment of pancreatic insufficiency in pancreatic cancer. Cancer 1983;52:346-52.
- 6. Partelli S, Frulloni L, Minniti C, Bassi C, Barugola G, D'Onofrio M, Crippa S, Falconi M. Faecal elastase-1 is an independent predictor of survival in advanced pancreatic cancer. Digestive and liver disease: official journal of the Italian Society of Gastroenterology and the Italian Association for the Study of the Liver 2012;44:945-51.
- 7. Sikkens EC, Cahen DL, de Wit J, Looman CW, van Eijck C, Bruno MJ. A prospective assessment of the natural course of the exocrine pancreatic function in patients with a pancreatic head tumor. Journal of clinical gastroenterology 2014;48:e43-6.
- 8. Dutta SK, Rubin J, Harvey J. Comparative evaluation of the therapeutic efficacy of a pH-sensitive enteric coated pancreatic enzyme preparation with conventional pancreatic enzyme therapy in the treatment of exocrine pancreatic insufficiency. Gastroenterology 1983;84:476-82.
- 9. Graham DY. An enteric-coated pancreatic enzyme preparation that works. Digestive diseases and sciences 1979;24:906-9.
- 10. Halgreen H, Pedersen NT, Worning H. Symptomatic effect of pancreatic enzyme therapy in patients with chronic pancreatitis. Scandinavian journal of gastroenterology 1986;21:104-8.
- 11. Valerio D, Whyte EH, Schlamm HT, Ruggiero JA, Blackburn GL. Clinical effectiveness of a pancreatic enzyme supplement. JPEN. Journal of parenteral and enteral nutrition 1981;5:110-4.
- 12. Lankisch PG, Lembcke B, Goke B, Creutzfeldt W. Therapy of pancreatogenic steatorrhoea: does acid protection of pancreatic enzymes offer any advantage? Zeitschrift für Gastroenterologie 1986;24:753-7.
- 13. Schneider MU, Knoll-Ruzicka ML, Domschke S, Heptner G, Domschke W. Pancreatic enzyme replacement therapy: comparative effects of conventional and enteric-coated microspheric pancreatin and acid-stable fungal enzyme preparations on steatorrhoea in chronic pancreatitis. Hepatogastroenterology 1985;32:97-102.
- 14. Delchier JC, Vidon N, Saint-Marc Girardin MF, Soule JC, Moulin C, Huchet B, Zylberberg P. Fate of orally ingested enzymes in pancreatic insufficiency: comparison of two pancreatic enzyme preparations. Alimentary pharmacology & therapeutics 1991;5:365-78.
- 15. Bruno MJ, Haverkort EB, Tijssen GP, Tytgat GN, van Leeuwen DJ. Placebo controlled trial of enteric coated pancreatin microsphere treatment in patients with unresectable cancer of the pancreatic head region. Gut 1998;42:92-6.

- 16. Dominguez-Muñoz JE, Nieto L, J. I-G. Pancreatic Enzyme Replacement Therapy and Nutritional Advice are Associated With Longer Survival in Patients With Unresectable Pancreatic Cancer Pancreas 2013;42:1347.
- 17. Fernandez-del Castillo CJ, Ramon E. Supportive care of the patient with advanced exocrine pancreatic cancer. UpToDate 2014.
- 18. Nouisa-Arvanitakis S, Stapleton FB, Linshaw MA, Kennedy J. Therapeutic approach to pancreatic extract-induced hyperuricosuria in cystic fibrosis. The Journal of pediatrics 1977;90:302-5.
- 19. Smyth RL, van Velzen D, Smyth AR, Lloyd DA, Heaf DP. Strictures of ascending colon in cystic fibrosis and high-strength pancreatic enzymes. Lancet 1994;343:85-6.
- 20. FitzSimmons SC, Burkhart GA, Borowitz D, Grand RJ, Hammerstrom T, Durie PR, Lloyd-Still JD, Lowenfels AB. High-dose pancreatic-enzyme supplements and fibrosing colonopathy in children with cystic fibrosis. The New England journal of medicine 1997;336:1283-9.
- 21. Gullo L, Pezzilli R, Gaiani S. Tolerability and safety of the long-term administration of pancreatic extracts. Pancreas 1997;14:210-2.
- 22. Seiler CM, Izbicki J, Varga-Szabo L, Czako L, Fiok J, Sperti C, Lerch MM, Pezzilli R, Vasileva G, Pap A, Varga M, Friess H. Randomised clinical trial: a 1-week, double-blind, placebo-controlled study of pancreatin 25 000 Ph. Eur. minimicrospheres (Creon 25000 MMS) for pancreatic exocrine insufficiency after pancreatic surgery, with a 1-year open-label extension. Alimentary pharmacology & therapeutics 2013;37:691-702.
- 23. Ramesh H, Reddy N, Bhatia S, Rajkumar JS, Bapaye A, Kini D, Kalla M, Thorat V. A 51-week, open-label clinical trial in India to assess the efficacy and safety of pancreatin 40000 enteric-coated minimicrospheres in patients with pancreatic exocrine insufficiency due to chronic pancreatitis. Pancreatology: official journal of the International Association of Pancreatology 2013;13:133-9.
- 24. Gubergrits N, Malecka-Panas E, Lehman GA, Vasileva G, Shen Y, Sander-Struckmeier S, Caras S, Whitcomb DC. A 6-month, open-label clinical trial of pancrelipase delayed-release capsules (Creon) in patients with exocrine pancreatic insufficiency due to chronic pancreatitis or pancreatic surgery. Alimentary pharmacology & therapeutics 2011;33:1152-61.